CLINICAL TRIAL: NCT07080385
Title: A Phase 2/3, Multicenter, Single-Arm, Open-Label Study Evaluating the Pharmacokinetics, Efficacy, and Safety of Encaleret in Pediatric Participants With Autosomal Dominant Hypocalcemia Type 1 (ADH1)
Brief Title: Pharmacokinetics, Efficacy, and Safety of Encaleret in Pediatric Participants With Autosomal Dominant Hypocalcemia Type 1 (ADH1)
Acronym: CALIBRATE-PEDS
Status: Recruiting | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Calcilytix Therapeutics, Inc., a BridgeBio company (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: CLTX-305-303
Record Dates: First submitted 2025-07-14; First posted 2025-07-23 (Actual); Last update posted 2026-01-14 (Actual); Status verified 2026-01

CONDITIONS: Autosomal Dominant Hypocalcemia Type 1 (ADH1)
Keywords: Autosomal dominant hypocalcemia type 1; ADH1; Encaleret

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Encaleret (Experimental): Participants will receive encaleret dosing in Period 1 (6 days), Period 2 (20 weeks) and Period 3 (4 weeks). Following completion of Period 3, participants will have the option to enter a long-term extension (LTE) to continue encaleret for an additional approximately 24 months or until the sponsor decides to end the study, whichever occurs first.
  Interventions: Drug: Encaleret

INTERVENTIONS:
Drug: Encaleret — Oral tablets, age-appropriate pediatric formulation (currently under development).

SUMMARY:
The overall objective of this study is to evaluate the pharmacokinetics (PK), efficacy, and safety of encaleret in pediatric participants from birth to 17 years of age with ADH1.

ELIGIBILITY:
Key Inclusion Criteria:

* Provide written informed consent (if legally permitted), or have written informed consent from a parent/legal guardian and provide assent (where required and as appropriate per local requirements)
* Have a documented pathogenic or likely pathogenic activating variant, or variant of uncertain significance of the calcium-sensing receptor (CASR), associated with biochemical findings of hypoparathyroidism at screening or a documented history of hypoparathyroidism as manifested by hypocalcemia and intact parathyroid hormone (PTH) <40 picogram per milliliter (pg/mL) (4.2 picomoles per liter [pmol/L])
* Have at least 1 symptom or sign of hypoparathyroidism at screening or a documented history of symptoms or signs of hypoparathyroidism
* Be on ADH1 treatment for at least 6 months before screening for cohorts 1 to 3, or for at least 3 months before screening for cohort 4

Key Exclusion Criteria:

* History of thyroid or parathyroid surgery
* History of renal transplantation
* History of cancer (except thyroid cancer, basal cell skin cancer, or squamous cell skin cancer), skeletal malignancies, bone metastases, irradiation (radiotherapy) to the skeleton, chemotherapy with alkylating agents, Paget disease, fibrous dysplasia, chronic osteomyelitis, bone infarcts, benign bone tumors with curettage and bone grafts, retinoblastoma, or Li-Fraumeni syndrome within 5 years before screening
* Received any investigational medicinal product within 30 days or 5 half-lives before Day 1, whichever is longer, or is in follow-up for another interventional clinical study during screening
* Treatment with a strong P-glycoprotein (P-gp) inhibitor within 300 days before screening for amiodarone or within 30 days before screening for any other strong P-gp inhibitor
* Treatment with cardiac glycosides, or is being breastfed while the participant's nursing mother is treated with cardiac glycosides, within 30 days before screening
* Presence or history of any disease or condition (eg, drug or alcohol dependence) that would affect the participant's safety, treatment compliance, or ability to complete the study, in the opinion of the investigator

Other protocol defined inclusion/exclusion criteria apply.

Ages: 0 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 28 (Estimated)
Dates: Start 2026-02-10 (Estimated); Primary Completion 2028-12 (Estimated); Study Completion 2030-12 (Estimated)

PRIMARY OUTCOMES:
Period 1: Maximum Plasma Concentration (Cmax) of Encaleret and Metabolites M1, and M3 | 5 days
Period 1: Area Under the Plasma Concentration-time Curve (AUC) of Encaleret and Metabolites M1, and M3 | 5 days
Period 3: Number of Participants with Albumin-corrected Blood Calcium (cCa) and Urinary Calcium (UCa) Excretion Response | Week 25

SECONDARY OUTCOMES:
Period 1: Change from Baseline in Blood cCa | Baseline up to Day 5
Period 1: Change from Baseline in Blood Intact Parathyroid Hormone (iPTH) Concentration | Baseline up to Day 5
Period 1: Change from Baseline in Blood Phosphate Concentration | Baseline up to Day 5
Period 1: Change from Baseline in Blood 1,25-(OH)2 Vitamin D Concentration | Baseline up to Day 5
Period 1: Change from Baseline in Blood Magnesium Concentration | Baseline up to Day 5
Period 1: Change from Baseline in 24-hour UCa in Toilet Trained Participants | Baseline up to Day 5
Period 1: Change from Baseline in Spot Ratio of UCa/Urinary Creatinine (UCr) In Non-toilet Trained Participants | Baseline up to Day 5
Period 3: Number of Participants with Blood iPTH Within the Reference Range | Week 25 (post-dose)
Period 3: Number of Participants with Blood Phosphate Within the Reference Range | Week 25
Period 3: Number of Participants with Blood Magnesium Within the Reference Range | Week 25
Period 3: Number of Participants with Blood 1,25-(OH)2 Vitamin D Within the Reference Range | Week 25
Periods 1, 2, and 3: Change from Baseline in Short Form-10 Health Survey for Children (SF-10) in Participants Aged ≥6 Years | Baseline up to Week 25
Periods 1, 2, and 3: Dose of Calcium Supplements and/or Active Vitamin D Analogs Used as Rescue Therapy | 25 weeks
Periods 1, 2, and 3: Dosing Frequency of Calcium Supplements and/or Active Vitamin D Analogs Used as Rescue Therapy | 25 weeks
Periods 1, 2, 3, and LTE: Number of Participants with Adverse Events (AEs) and Serious AEs (SAEs) | 145 weeks
LTE: Change from Baseline in Blood cCa | Baseline up to 145 weeks
LTE: Change from Baseline in Blood iPTH Concentration | Baseline up to 145 weeks
LTE: Change from Baseline in Blood Phosphate Concentration | Baseline up to 145 weeks
LTE: Change from Baseline in Blood 1,25-(OH)2 Vitamin D Concentration | Baseline up to 145 weeks
LTE: Change from Baseline in Blood Magnesium Concentration | Baseline up to 145 weeks
LTE: Change from Baseline in 24-hour UCa In Toilet Trained Participants | Baseline up to 145 weeks
LTE: Change from Baseline in Spot Ratio of UCa/UCr In Non-toilet Trained Participants | Baseline up to 145 weeks
LTE: Change from Baseline in SF-10 in Participants Aged ≥6 Years | Baseline up to 145 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Calcilytix Medical Director, Study Director — Calcilytix Therapeutics, Inc., a BridgeBio company
Locations (1):
- The Children's Hospital of Philadelphia, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No